CLINICAL TRIAL: NCT00005553
Title: Prospective Assessment After Pediatric Cardiac Ablation (PAPCA)
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5097; R01HL058620 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2005-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Arrhythmia; Tachycardia, Supraventicular
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Arrhythmias, Cardiac; Tachycardia | interventions — Catheter Ablation

INTERVENTIONS:
Procedure: Catheter Ablation

SUMMARY:
To evaluate children undergoing catheter ablation at pediatric centers in North America in order to provide information on the incidence rate of serious cardiac damage as a result of ablation, the incidence rate and time course of recurrence after initially successful ablation, and the incidence rate of proarrhythmia following ablation.

DETAILED DESCRIPTION:
BACKGROUND:

Radiofrequency catheter ablation is a catheterization laboratory technique for the cure of cardiac arrhythmias, which has become common in pediatric cardiology practice. Recent analyses have suggested that ablation therapy is more cost-effective compared not only with surgery, but also with antiarrhythmic medication. Despite a good initial success rate of the technique, and a low initial complication rate, there is concern about possible long-term effects with the technique in the pediatric age group. There are reports not only of damage to cardiac valves, but also the development of new arrhythmias, including sudden death, as a result of ablations in children. Recurrences are observed frequently following initially successful procedures. Finally, there are animal data to suggest that immature myocardium is more prone to severe damage as a result of ablation procedures. Few, if any, data exist to support the long-term safety of these ablation techniques in children. Therefore, before ablation therapy becomes the standard approach in children, it is important to carefully assess the long-term risks in this patient group.

DESIGN NARRATIVE:

Multi-center, prospective, five-year study. The collection of these data was intended to provide the following information: 1) the incidence of serious cardiac damage as a result of ablation; 2) the incidence and time course of recurrence after initially successful ablation; and 3) the incidence of proarrhythmia following ablation. A total of 480 pediatric patients were enrolled prospectively and evaluated both before ablation of supraventricular tachycardia and at intervals following ablation with clinical history and examination, electrocardiogram, 24-hour Holter monitor, and echocardiogram, with non-invasive studies read by outside consultants. In addition, a complete Registry of pediatric patients undergoing ablation at the participating centers was established to allow comparisons with the study group and to provide population estimates of success and complication rates.

ELIGIBILITY:
No eligibility criteria

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1998-05; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: George Van Hare — Stanford University

REFERENCES:
- [Background] Van Hare GF, Carmelli D, Smith WM, Kugler J, Silka M, Friedman R, Atkins D, Saul P, Schaffer M, Byrum C, Dunnigan A, Colan S, Serwer G; Pediatric Electrophysiology Society. Prospective assessment after pediatric cardiac ablation: design and implementation of the multicenter study. Pacing Clin Electrophysiol. 2002 Mar;25(3):332-41. doi: 10.1046/j.1460-9592.2002.00332.x. PMID 11990663
- [Background] Van Hare GF, Javitz H, Carmelli D, Saul JP, Tanel RE, Fischbach PS, Kanter RJ, Schaffer M, Dunnigan A, Colan S, Serwer G; Pediatric Electrophysiology Society. Prospective assessment after pediatric cardiac ablation: demographics, medical profiles, and initial outcomes. J Cardiovasc Electrophysiol. 2004 Jul;15(7):759-70. doi: 10.1046/j.1540-8167.2004.03645.x. PMID 15250858
- [Background] Van Hare GF, Javitz H, Carmelli D, Saul JP, Tanel RE, Fischbach PS, Kanter RJ, Schaffer M, Dunnigan A, Colan S, Serwer G; Participating Members of the Pediatric Electrophysiology Society. Prospective assessment after pediatric cardiac ablation: recurrence at 1 year after initially successful ablation of supraventricular tachycardia. Heart Rhythm. 2004 Jul;1(2):188-96. doi: 10.1016/j.hrthm.2004.03.067. PMID 15851152
- [Background] Anand RG, Rosenthal GL, Van Hare GF, Snyder CS. Is the mechanism of supraventricular tachycardia in pediatrics influenced by age, gender or ethnicity? Congenit Heart Dis. 2009 Nov-Dec;4(6):464-8. doi: 10.1111/j.1747-0803.2009.00336.x. PMID 19925541